CLINICAL TRIAL: NCT02137655
Title: Prospective Descripive Study of Subacute Function After Total Hip or Knee Arthroplasty
Brief Title: Recovery After Fast Track THA / TKA
Acronym: 0-21
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Eske Kvanner Aasvang, MD, DMSci, Rigshospitalet, Denmark
Other Study IDs: H-3-2014-005
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Hip and Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The development and implementation of "fast-track" principles in total knee and hip arthroplasty have resulted in early recovery and rehabilitation alongside a reduced length of hospital stay. This without a concomitant increase in morbidity or readmissions for medical or surgical complications and with reduced mortality. However, only little is known about function in the subacute period after arthroplasty, and there is a need for further data on physical and psychological functioning following discharge from hospital.This to ensure, that the positive results from the perioperative setting are carried forward in the subacute phase.

DETAILED DESCRIPTION:
Data will be published in three papers:

1. "Physical function and related factors following discharge from THA and TKA" Luna IE, Kehlet H, Aasvang EK.
2. "Postoperative hypoxemia following fast-track hip and knee arthroplasty" Luna IE, Kehlet H, Aasvang EK.
3. "Cognitive dysfunction after fast-track hip- and knee arthroplasty - prevalence and related factors". Luna IE, Kehlet H, Aasvang EK.

ELIGIBILITY:
Inclusion Criteria:

* Primary total hip or knee arthroplasty
* Age 55 to 80 years

Exclusion Criteria:

* Deficient written or spoken danish
* Alcohol abuse (>21 U per week)
* Immunocompromised
* Anticoagulant therapy
* ASA class 4-5
* Functional impairment from psychological or neurological disease
* Sleepapnea

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hip or knee osteoarthritis referred for total joint arthroplasty.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2014-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Pain | 48 hours postoperatively
  VAS when walking

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Gentofte hospital, Gentofte Municipality, Capital Region
  - Vejle Sygehus, Vejle, Region Syd